CLINICAL TRIAL: NCT02338050
Title: A Phase II Study of the Anti-CD22 Recombinant Immunotoxin Moxetumomab Pasudotox (CAT-8015, HA22) in Children With B-lineage Acute Lymphoblastic Leukemia and Minimal Residual Disease Prior to Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Moxetumomab Pasudotox (CAT-8015, HA22) in Children With B-lineage Acute Lymphoblastic Leukemia and Minimal Residual Disease Prior to Allogeneic Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other); Pediatric Blood and Marrow Transplant Consortium (Other); MedImmune LLC (Industry); St. Baldrick's Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-MOXE
Record Dates: First submitted 2015-01-06; First posted 2015-01-14 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
Keywords: ALL; Moxetumomab Pasudotox; Moxe; CAT-8015, HA22
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — immunotoxin HA22; HA 22

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Moxetumomab Pasudotox (Experimental): Moxetumomab pasudotox 32 mcg/kg/dose IV every other day for a total of 6 doses. Dexamethasone 2.5 mg/m2/dose (or corticosteroid equivalent) will be administered before and after each dose of moxetumomab pasudotox.
  Interventions: Biological: Moxetumomab Pasudotox

INTERVENTIONS:
Biological: Moxetumomab Pasudotox
  Other Names: (CAT-8015, HA22)

SUMMARY:
This is a phase II, open-label, nonrandomized, prospective study to evaluate the activity, safety, and feasibility of administration of moxetumomab pasudotox in the pre-allogeneic hematopoietic cell transplantation (HCT) setting to patients with B-lineage Acute Lymphoblastic Leukemia (ALL) who are in a morphologic complete remission and have pre-transplant minimal residual disease (MRD) > 0.01% (detected by flow cytometry). The primary objective of this study is to determine if treatment with moxetumomab pasudotox in the MRD positive setting is able to lead to MRD negativity (< 0.01% by flow cytometry) or at least a 1-log10 reduction in MRD prior to allogeneic HCT.

DETAILED DESCRIPTION:
This is a Phase 2 study designed to assess safety, feasibility and clinical activity of pre-HCT moxetumomab pasudotox for patients with ALL in morphologic CR but with MRD. It is hypothesized that subjects in a morphologic complete remission with proven minimal residual disease (MRD) after chemotherapy for ALL planned for allogeneic HCT who receive a course of moxetumomab pasudotox prior to the start of conditioning will show a marked reduction or elimination of detectable MRD after moxetumomab pasudotox treatment without adverse impact on the feasibility or safety of allogeneic HCT.

The primary objective of this study is to determine if treatment with moxetumomab pasudotox in the MRD positive setting is able to lead to MRD negativity (< 0.01% by flow cytometry) or at least a 1-log10 reduction in MRD prior to allogeneic HCT.

Secondary objectives to be studied include: toxicity profile (including safety and feasibility of administration in the pre-HCT setting and ability to proceed to transplant, incidence of capillary leak syndrome, hemolytic uremic syndrome and other post-HCT toxicities), comparison of quantitative MRD assessments, progression-free survival, overall survival, pharmacokinetic profiles, immunogenicity to moxetumomab pasudotox, transplant-related mortality, acute and chronic graft-versus-host disease (GVHD), and relapse.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 6 months and < 25 years of age
2. Histologically confirmed diagnosis of B-lineage ALL. Verification of CD22 expression is not required
3. Bone marrow in morphologic remission (any remission number) defined as < 5% blasts (M1 classification) performed in local institution lab
4. CNS 1 (< 5/μL WBCs in CSF and cytospin negative for blasts)
5. Evidence of bone marrow MRD defined as ≥ 0.01% by flow cytometry performed in the study central lab
6. Candidate committed to HCT independent of participation in this study, with the following requirements:

   * Meets local transplant center eligibility requirements for HCT
   * In the opinion of the HCT center will be ready to begin pre-transplant conditioning within 6 weeks of trial enrollment from a medical and psychosocial standpoint
   * Has an available HCT donor or identified cord blood unit. Related and unrelated donors, and bone marrow, peripheral blood, or cord blood stem cell sources allowed
7. Adequate organ function including the following:

   * Hepatic function: Total bilirubin < 1.5 × upper limit of normal (ULN) (except in the case of subjects with known Gilbert's disease: < 5 × ULN) and transaminases (alanine aminotransferase (ALT) and aspartate aminotransferase (AST)) < 3 × ULN based on age- and institution specific laboratory-specific normal ranges
   * Renal function: Age-adjusted normal serum creatinine is required. A 24-hour creatinine clearance value > 60 mL/min/1.73 m2 (updated Schwartz formula or nuclear GFR) must be obtained if serum creatinine is elevated.
   * Hematologic function: Absolute neutrophil count (ANC) > 500/μL and platelet count > 25,000/μL without transfusion
   * Oxygen saturation at rest or with exercise > 88% as measured by pulse oximeter or PaO2 > 55 mm Hg without need for supplemental oxygen at rest or with activity
   * Serum albumin > 2 g/dL
8. Performance status:

   * Subjects ≥ 16 years of age: Karnofsky ≥ 60% (Appendix A)
   * Subjects < 16 years of age: Lansky scale ≥ 60% (Appendix A)
   * Subjects who are unable to walk because of paralysis, but who are upright in a wheel chair will be considered ambulatory for the purpose of calculating the performance score
9. Patients > 18 years of age must have the ability to give informed consent according to applicable regulatory and local institutional requirements. Legal guardian permission must be obtained for patients < 18 years of age. Pediatric patients will be included in age appropriate discussion in order to obtain assent
10. Sexually active female subjects of childbearing potential and male subjects and their sexual partners who are of childbearing potential must agree to use contraception

Exclusion Criteria:

1. Active extramedullary disease at any site. (Note: Definitive therapy of known previous sites of extramedullary disease is allowed)
2. Females who are breast-feeding or pregnant
3. Subjects with known 11q23 MLL rearrangement are excluded.
4. Prior therapy:

   * Prior treatment with CAT-3888 (BL22), moxetumomab pasudotox (CAT-8015, HA22), any pseudomonas-exotoxin-containing compound, or any anti-CD22 directed therapy at any time in the past
   * Prior allogeneic or autologous HCT or adoptive cellular therapies, including T-cell chimeric antigen receptor (CAR) therapy
   * Chemotherapy < 2 weeks prior to starting study drug with the following exception: There is no time restriction in regard to prior intrathecal chemotherapy provided there is complete recovery from any acute toxic effects of such
   * Monoclonal antibody therapy < 30 days from study enrollment
   * Other investigational agents currently or within 30 days prior to study enrollment
5. Subjects with an absolute contraindication to corticosteroid administration
6. HIV infection (due to increased risk of severe infection and unknown interaction of moxetumomab pasudotox with antiretroviral drugs)
7. Active hepatitis B or C infection as defined by seropositivity for hepatitis B (hepatitis B surface antigen [HbsAg]) or hepatitis C (hepatitis C antibody) and elevated liver transaminases (defined as above the ULN per the institution normal ranges)
8. Second malignancy other than non-basal cell carcinoma of the skin or in situ carcinoma of the cervix, unless the tumor was treated with curative intent at least two years previously and subject is in remission
9. Subject with clinical or laboratory evidence of active DIC
10. Subject with prior history of thrombotic microangiopathy or HUS within 3 months prior to enrollment
11. History of known congenital hypercoagulable condition
12. Previous life-threatening anaphylactic reactions to prior monoclonal antibody-based immunotherapy or any component of the moxetumomab pasudotox formulation
13. Subjects who will be or are currently being treated with high dose estrogen (high dose is defined as >0.625mg daily as conjugated estrogens or equivalent) within 7 days prior to study enrollment

Ages: 6 Months to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
MRD negativity | change in MRD levels between baseline and 3-10 days post last Moxe dose
  The primary endpoint is the event of whether patients successfully achieved either MRD negativity (defined as <0.01%) or at least 1 log10 reduction in MRD levels using flow cytometry via central laboratory testing after moxetumomab treatment but prior to HCT relative to pre-moxetumomab MRD measurement (baseline). The proportion of patients who become MRD negative or who have at least a 1-log10 reduction from baseline will be summarized and 80% confidence intervals will provided. An exploratory analysis of the association between CD22 expression at eligibility and the response rate will also be conducted.

SECONDARY OUTCOMES:
MRD level and its log reduction from baseline | baseline and 3-10 days post last Moxe dose
  will be described quantitatively at each time point using median and range. Values that go below the lower limit of detection (<0.01%) will be set to the lower limit to obtain a conservative estimate of the log reduction. A test of whether the MRD levels are significantly reduced relative to baseline will be conducted using the Wilcoxon signed rank test. Agreement between quantitative MRD assessments using flow cytometry and molecular sequencing (immunosequencing) will be assessed using reliability coefficients and Bland-Altman plots, applied to the log transformed MRD levels. The correlation between CD22 expression at eligibility and log reduction in MRD from baseline will be described using Spearman's rank correlation.
Overall Survival (OS) | from Moxe Dose 1 through date of death from any cause (assessed through 2 years post HCT or last Moxe dose)
  is defined as the time from the start of treatment with moxetumomab pasudotox until death for the treated population. The OS will be censored if the patient did not die at the end of the study. For transplant population, the start time is from the date of transplant. Kaplan-Meier estimator will be used for the median or survival rate at a particular time.
Progression-free survival (PFS) | from Moxe Dose 1 through date of progression or death from any cause (assessed through 2 years post HCT or last Moxe dose)
  is defined as the time from the start of treatment with moxetumomab pasudotox until the documentation of disease progression or death due to any cause, whichever occurs first, for the treated population. PFS will be censored if the patient did not relapse by the last visit. For transplant population, the start time is from the date of transplant. Kaplan-Meier estimator will be used for the median or survival rate at a particular time.
Proportion of patients proceeding to transplant | from Moxe Dose 1 through Day 0 of transplant
  will be described, along with a breakdown of the reasons for not proceeding to transplant and their frequencies.
Relapse | from Moxe Dose 1 through date of relapse (assessed through 2 years post HCT or last Moxe dose)
  Relapse will be defined by the presence of > 5% bone marrow blasts by morphology on an aspirate sample, or by evidence of peripheral blasts or extramedullary disease. The proportion of relapse will be summarized for both the treated population (from start of treatment) and transplant population (from date of transplant), using the cumulative incidence estimator with death in the absence of relapse as the competing event.
Transplant-related mortality (TRM) | from Day 0 of transplant through date of death without evidence of disease progression or recurrence (assessed through 2 years post HCT)
  An event for this endpoint is death without evidence of disease progression or recurrence. TRM will be summarized using cumulative incidence for transplant population.
Acute GVHD | from Day 0 of transplant through first onset date of acute GVHD grades II-IV and grades III-IV (assessed through 2 years post HCT)
  The events are the incidences of grades II-IV and grades III-IV acute GVHD from day of transplant. The first day of acute GVHD onset at a certain grade will be used to calculate a cumulative incidence curve for that acute GVHD grade. Death is considered as a competing risk. Transplant population will be used.
Chronic GVHD | from Day 0 of transplant through first onset date of chronic GVHD (assessed through 2 years post HCT)
  The cumulative incidence of chronic GVHD starting at the day of transplant will be summarized, treating death as a competing risk. Transplant population will be used.
Clinical Laboratory Values | from baseline through 3-10 days post last Moxe dose
  The values and abnormalities for relevant laboratory tests will be summarized by descriptive statistics (e.g., number of subjects, mean, standard deviation, median, minimum, maximum, proportions, etc.) at each time point and also for change from baseline value. Baseline will be defined as the last non-missing value prior to treatment with moxetumomab pasudotox.
Pre-transplant toxicities: Pre-transplant adverse events | from Moxe Dose 1 through 30 days after the last dose of study drug or until start of conditioning regimen
  Pre-transplant adverse events will be collected until 30 days after the last dose of study drug or until transplant and will be tabulated by severity and relationship to the study drug. Post-transplant adverse events will be analyzed separately as described in the next section.
  Capillary Leak Syndrome, hemolytic uremic syndrome, ocular toxicities and cytokine release syndrome/infusional reactions, as well as death which is possibly, probably or definitely related to moxetumomab pasudotox are Adverse Events of Interest and will be further analyzed by examining their correlation with other clinical variables.
Post-Transplant Toxicities: Unexpected SAEs | start of conditioning regimen and continuing for 60 days from Day 0 of transplant
  Unexpected SAEs will be tabulated by severity and relationship to study drug. The cumulative incidence of thrombotic microangiopathy (TMA), and hepatic veno-occlusive disease (VOD) will be described in transplanted patients, treating death as a competing risk. Transplanted population will be used for these analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Wayne, MD, Study Chair — Children's Hospital Los Angeles; Nirali N Shah, MD, Study Chair — National Institutes of Health (NIH)
Locations (4):
- United States (4):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Shah NN, Schneiderman J, Kuruvilla D, Bhojwani D, Fry TJ, Martin PL, Schultz KR, Silverman LB, Whitlock JA, Wood B, Vainshtein I, Adams A, Confer D, Pulsipher MA, Chaudhury S, Wayne AS. Fatal capillary leak syndrome in a child with acute lymphoblastic leukemia treated with moxetumomab pasudotox for pre-transplant minimal residual disease reduction. Pediatr Blood Cancer. 2021 Jan;68(1):e28574. doi: 10.1002/pbc.28574. Epub 2020 Sep 22. No abstract available. PMID 32959985